CLINICAL TRIAL: NCT03312452
Title: The Role of Infusion Pumps in Preventing the Over-Administration of Intravenous Fluid in Pediatric Dental Surgeries
Brief Title: The Incidence of IV Fluid Over-administration in Pediatric Dental Surgeries When Infusion Pumps Are Employed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Jonathan Gamble, Assistant Professor, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DBJG17-165
Record Dates: First submitted 2017-10-12; First posted 2017-10-17 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Dental Caries
Keywords: Pediatric; Perioperative; Intravenous fluid
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will blinded to group allocation by concealment of the IV fluid delivery device in the operating room. Analysts will be presented with data that has been coded to conceal each participants' allocation to either the intervention or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infusion pump group (Experimental): Study subjects assigned to this group will receive intravenous fluid via an infusion pump (Hospira plum pump) during their surgery.
  Interventions: Device: Hospira plum pump
- Gravity drip group (Active Comparator): Study subjects assigned to this group will receive intravenous fluid via a gravity drip device during their surgery.
  Interventions: Device: Gravity drip device

INTERVENTIONS:
Device: Hospira plum pump — The Hospira plum pump enables the clinician to program a specific volume of intravenous fluid and define a period of time over which to administer this fluid.
  Arms: Infusion pump group
Device: Gravity drip device — Study subjects assigned to this group will receive intravenous fluid via a gravity drip device during their surgery.
  Arms: Gravity drip group

SUMMARY:
A prospective, analyst-blinded, randomized control trial to assess the incidence of intravenous (IV) fluid over-administration in the setting of pediatric dental surgeries. Anesthetists will be randomized to either administer their IV fluid through an infusion pump or a gravity drip device.

DETAILED DESCRIPTION:
In the perioperative setting, IV fluids are administered to mitigate the effects of preoperative fasting and sources of fluid loss that are unique to surgical intervention. Significant harms have been associated with the over-administration of IV fluid in pediatric patients. Infusion pumps have been shown to reduce medication administration errors in inpatients receiving continuous IV infusions. In contrast, laboratory experiments have demonstrated that gravity driven fluid delivery systems are influenced by numerous extrinsic factors. To date, no work has investigated the perioperative incidence of IV fluid over-administration in pediatric patients randomized either to infusion pumps (intervention) or gravity-fed IV systems (control).

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 and 2 children presenting for dental surgery

Exclusion Criteria:

* Children with pre-existing cardiac, renal, pulmonary or endocrine disease. In addition any child with an ASA score of 3 or greater.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 103 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-10-19 (Actual); Study Completion 2018-10-19 (Actual)

PRIMARY OUTCOMES:
Average absolute difference between volume prescribed and infused | From initiation of intravenous until arrival in the recovery room, up to three hours
  Difference in volume originally prescribed and ultimately administered

SECONDARY OUTCOMES:
Volume of intravenous fluid administered | From initiation of intravenous until arrival in the recovery room, up to three hours
  Volume of fluid received over surgical course (mL/kg/hr)
Average percent difference between volume prescribed and infused | From initiation of intravenous until arrival in the recovery room, up to three hours
  Percent difference in volume originally prescribed and ultimately administered

CONTACTS AND LOCATIONS:
Overall Officials: Duncan EJ Bowes, M.D., Principal Investigator — Resident principal investigator
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bowes DE, Gamble JJ, Bajwa JS. Using automated pump-delivery devices to reduce the incidence of excessive fluid administration during pediatric dental surgery: a randomized-controlled trial. Can J Anaesth. 2020 Nov;67(11):1535-1540. doi: 10.1007/s12630-020-01776-4. Epub 2020 Aug 5. PMID 32761316